CLINICAL TRIAL: NCT03953846
Title: A Long-term Non-interventional Registry Study to Assess the Effectiveness and Safety of the NUsurface® Meniscus Implant
Brief Title: NUsurface Implant Registry
Acronym: NIR
Status: Terminated | Type: Observational
Why Stopped: Active Implants Europe closed operations
Sponsor: Active Implants (Industry)
Responsible Party: Sponsor
Other Study IDs: 01003
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-04

CONDITIONS: Meniscus; Degeneration; Knee Osteoarthritis; Knee Pain Chronic
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this active post-market surveillance clinical registry study is to further characterize the therapeutic effect, the long-term safety and effectiveness of the NUsurface® meniscus implant in the real-world post-marketing setting

DETAILED DESCRIPTION:
Patients eligible for the Registry includes any patient who received or is scheduled to receive the NUsurface® meniscus implant and meets the Registry inclusion criteria (Evidence of a personally signed and dated informed consent document). The NUsurface Implant Regitstry is about data collection only and under routine standard of care by treating physician. Data collection points are pre-op (i.e. baseline), surgery and multiple times after surgery during the first 6 months to correspond to clinic standard of care schedules, 6 months, 1 year post-operatively and then yearly thereafter out to 10 years.Surveys used are KOOS; Knee injury and Osteoarthritis Outcome Score & WOMET; Western Ontario Meniscal Evaluation Tool.

ELIGIBILITY:
Inclusion Criteria:

* New or current treatment with the NUsurface® meniscus implant
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the Registry.

Exclusion Criteria:

* There are no protocol exclusion criteria; all subjects who meet the inclusion criteria are eligible for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population eligible for this protocol includes any subject who received or is scheduled to receive the NUsurface® meniscus implant and meets the Registry inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
KOOS (Knee Osteoarthritis Outcome Score) Pain improvement | 24 months
  a responder is defined as a patient with an increase of at least 20 points on the KOOS pain assessment
WOMET (Western Ontario Meniscus Evaluation Tool) score improvement | 24 months
  a responder is defined as a patient with an increase of at least 12 points on the WOMET assessment

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Threharne, PhD, Study Director — Active Implants LLC
Locations (6):
- AZ Monica vzw, Deurne, Belgium
- Germany (3):
  - Sporthopaedicum, Berlin
  - University of Brandenburg, Brandenburg
  - Klinikum der Universität München, München
- Shamir Medical Center, Ẕerifin, Israel
- Maastricht UMC, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided